CLINICAL TRIAL: NCT01095068
Title: Beneficial Effects of Exercise Training on Physical Capacity in Type 2 Diabetics: Improvement in Skeletal Muscle Energetic Capacity, Endothelial Dysfunction and Glycemic Control
Brief Title: Effects of Physical Exercise in Type 2 Diabetics
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3661
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- physical exercise (Experimental): Physical exercise
  Interventions: Behavioral: Physical exercise

INTERVENTIONS:
Behavioral: Physical exercise

SUMMARY:
The aim of this study is to evaluate the improvement in skeletal muscle energetic capacity, endothelial dysfunction and glycemic control induced by physical training in 20 sedentary patients with a type 2 diabetes.The protocol consists in a physical training program with 3 sessions of 30 minutes per week during six consecutive weeks. A skeletal muscle biopsy, a cardiac and humeral artery ultrasounds, a glycemic and tensional holters will be performed before and at the end of the physical training program.

ELIGIBILITY:
Inclusion Criteria:

* sedentary adult with type 2 diabetes
* BMI between 25 and 35 kg/m²
* Hba1c < 10 %

Exclusion Criteria:

* unstable coronary artery disease
* advanced peripheral occlusive arterial disease
* proteinuria > 3 g/d and / or creatinine clearance < 30 ml / mn
* advanced diabetic neuropathy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain PRADIGNAC, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (3):
- France (3):
  - Médecine Interne et Nutrition, Hôpital Civil, Hôpitaux universitaires de Strasbourg, Strasbourg
  - Service de Physiologie et d'Explorations Fonctionnelles, Nouvel Hôpital Civil, Hôpitaux universitaires de Strasbourg, Strasbourg
  - Service de Médecine Interne et Nutrition, Hôpital de Hautepierre, Hôpitaux universitaires de Strasbourg, Strasbourg